CLINICAL TRIAL: NCT07393516
Title: EFFECTS OF VARIABLE-PRIORITY DUAL-TASK TRAINING ON BALANCE, GAIT, AND QUALITY OF LIFE IN ELDERLY WOMEN IN CHINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu Xiao (Other)
Responsible Party: Sponsor-Investigator, Yu Xiao, Phd, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JKEUPM-2023-373
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Dual-task; Older Adults (65 Years and Older); Older Adults, Balance; Balance; Gait; Quality of Life (QOL)
Keywords: Balance; Gait; Older adults; Quality of life; dual-task training; Variable-priority dual-task training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Variable-priority dual-task training (Experimental): Variable priority dual-task training requires participants to perform cognitive-motor dual-task training while adjusting attention priorities based on instructions such as "posture priority" or "cognitive priority." During training, the coach monitored behaviour for adherence to the instructed priority (e.g., excessive stopping to respond during cognitive-priority bouts, reduced responding/ignoring prompts during cognitive-priority bouts, or unsafe postural behaviour during posture-priority bouts). When deviations were observed, standardized corrective prompts were delivered immediately and the priority instruction was restated. Cognitive-task performance (correct/total responses) was recorded for each bout as an adherence indicator of engagement with the instructed attentional priority. Marked accuracy deterioration or obvious non-compliance triggered real-time coaching prompts to restore the intended priority strategy while maintaining safe postural control.
  Interventions: Behavioral: Variable-Priority Cognitive-Motor Dual-Task Training
- Fixed-priority dual-task training (Active Comparator): Fixed-priority dual-task training requires participants to perform cognitive-motor dual-task training simultaneously. At the beginning of each session and before each motor-task set, participants were instructed to "pay equal attention to the motor and cognitive tasks throughout," aiming to maintain safe, stable movement while responding as accurately as possible. Participants were asked to repeat the instruction in their own words to confirm understanding. During training, the coach monitored behaviour for signs of disproportionate prioritization (e.g., pausing the motor task to answer, ignoring the cognitive prompt, or unsafe postural behaviour). Standardized reminders (e.g., "keep both tasks equally important") were delivered when needed. Cognitive responses were checked in real time, and incorrect responses were corrected immediately to reinforce engagement with the cognitive task while maintaining safe postural control.
  Interventions: Behavioral: Fixed-Priority Cognitive-Motor Dual-Task Training
- Phsical training (Active Comparator): The PT group first performed a 10-minute warm-up exercise. Then, in the order of the exercise tasks, they performed sit-ups, stand-ups, seated rowing, object transfer, obstacle avoidance, and connected walking training. Finally, a 10-minute relaxation activity was performed. Session duration, weekly frequency, and supervision were matched across the VPDT and FPDT groups, but PT consisted only of single-task exercises (no cognitive tasks or priority instructions).
  Interventions: Behavioral: Phsical training

INTERVENTIONS:
Behavioral: Variable-Priority Cognitive-Motor Dual-Task Training — Intervention Description (VPDT):
  Participants will receive variable-priority cognitive-motor dual-task training (VPDT) for 12 weeks. Training will be delivered in supervised sessions 3 times/week, 60 minutes/session, in a small group format. Each session combines functional balance and gait tasks (e.g., sit-to-stand, obstacle negotiation, line walking, turning, transfers) with concurrent cognitive tasks (e.g., serial subtraction/1-back/semantic fluency). Variable-priority instructions are used: participants are coached to flexibly shift attention between the motor and cognitive task across repetitions/blocks, with individualized cueing. Attendance is recorded each session; adverse events are monitored and managed according to a predefined safety protocol.
  Arms: Variable-priority dual-task training
Behavioral: Fixed-Priority Cognitive-Motor Dual-Task Training — Intervention Description (FPDT):
  Participants will receive fixed-priority cognitive-motor dual-task training (FPDT) for 12 weeks, supervised 3 times/week, 60 minutes/session. The motor tasks and cognitive tasks are matched to the VPDT group in type and total practice time. Fixed-priority instructions are used: participants are instructed to maintain equal and consistent attention to both tasks simultaneously throughout training, without shifting priorities across blocks. Progression and safety monitoring follow the same principles as VPDT. Attendance and adverse events are documented.
  Arms: Fixed-priority dual-task training
Behavioral: Phsical training — The PT group first performed a 10-minute warm-up exercise. Then, in the order of the exercise tasks, they performed sit-ups, stand-ups, seated rowing, object transfer, obstacle avoidance, and connected walking training. Finally, a 10-minute relaxation activity was performed. Session duration, weekly frequency, and supervision were matched across the VPDT and FPDT groups, but PT consisted only of single-task exercises (no cognitive tasks or priority instructions).
  Arms: Phsical training

SUMMARY:
This clinical trial aims to investigate the effects of variable-priority dual-task training on balance, gait, and quality of life in Chinese elderly women, exploring more effective training methods to help healthy elderly women improve balance and gait performance, reduce fall rates, and enhance quality of life. The trial primarily seeks to address the following questions:

H01: Between the three intervention groups (VPDT, FPDT, and PT), there are no statistically significant differences in balance among healthy older Chinese women at baseline (T1), week 6 (T2), or week 12 (T3).

H02: Between the three intervention groups (VPDT, FPDT, and PT), there are no statistically significant differences in gait among healthy older Chinese women at baseline (T1), week 6 (T2), or week 12 (T3).

H03: Between the three intervention groups (VPDT, FPDT, and PT), there are no statistically significant differences in QoL among healthy older Chinese women at baseline (T1), week 6 (T2), or week 12 (T3).

Researchers will compare variable-priority dual-task training with a placebo (fixed-priority dual-task training and physical training) to determine whether variable-priority dual-task training effectively improves balance, gait, and quality of life in Chinese elderly women.

Participants will:

Undergo three 60-minute training sessions per week for 12 weeks; Each session combines concurrent cognitive and physical training, with slight variations in content across the three groups; Outcome measurements will be taken at baseline, week 6 post-intervention, and week 12 post-intervention.

ELIGIBILITY:
Inclusion Criteria:

(1) age ≥65 years; (2) no severe visual or hearing impairments; (3) no limb disabilities or physical mobility impairments, able to stand and walk independently without the use of walking aids; (4) no neurological diseases or cognitive impairment; (5) MoCA score ≥26; (6) informed consent and voluntary participation.

Exclusion Criteria:

(1) severe cardiovascular, pulmonary, or musculoskeletal system diseases; (2) neurological diseases severely affecting balance function, such as stroke or Parkinson's disease; (3) mental illnesses such as depression or use of psychiatric medications; (4) need for assistive devices for walking; (5) simultaneous participation in other clinical trials.

Ages: 65 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 75 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Dual-Task 10-Meter Walk Test | From enrollment to the end of treatment at 12 weeks
10-Meter Walk Test | From enrollment to the end of treatment at 12 weeks
Timed Up and Go Test | From enrollment to the end of treatment at 12 weeks
Dual-Task Timed Up and Go Test | From enrollment to the end of treatment at 12 weeks
Five Times Sit-to-Stand Test | From enrollment to the end of treatment at 12 weeks
Single-Legged Closed-Eyed Standing Test | From enrollment to the end of treatment at 12 weeks
Berg Balance Scale | From enrollment to the end of treatment at 12 weeks
Activities-Specific Balance Confidence Scale | From enrollment to the end of treatment at 12 weeks

SECONDARY OUTCOMES:
36-Item Short Form of Health Survey | From enrollment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Jinheyuan Community Senior Citizens Activity Center, Hongshan District, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share individual participant data (IPD) has not yet been determined. The study team is developing a data management and sharing plan and will consider data sharing after study completion, subject to ethics approval, participant consent, and institutional policies. Any shared dataset would be de-identified and provided under appropriate data-use agreements.

REFERENCES:
- [Result] Trombini-Souza F, de Maio Nascimento M, da Silva TFA, de Araujo RC, Perracini MR, Sacco ICN. Dual-task training with progression from variable- to fixed-priority instructions versus dual-task training with variable-priority on gait speed in community-dwelling older adults: A protocol for a randomized controlled trial : Variable- and fixed-priority dual-task for older adults. BMC Geriatr. 2020 Feb 22;20(1):76. doi: 10.1186/s12877-020-1479-2. PMID 32087694
- [Result] Effect of agility training under single-task condition versus training under dual-task condition with different task priorities to improve balance in the elderly.
- [Result] Lussier M, Bugaiska A, Bherer L. Specific transfer effects following variable priority dual-task training in older adults. Restor Neurol Neurosci. 2017;35(2):237-250. doi: 10.3233/RNN-150581. PMID 27372514
- [Result] Gavzer K. How do employees feel about working in a veterinary practice? J Am Vet Med Assoc. 1989 Jul 15;195(2):182-3. No abstract available. PMID 2768031
- [Result] Gutschik E. Experimental endocarditis in rabbits. 6. Results of long-term combined therapy of Streptococcus faecalis endocarditis with penicillin and streptomycin. Acta Pathol Microbiol Immunol Scand B. 1982 Feb;90(1):37-47. PMID 6805250